CLINICAL TRIAL: NCT04539639
Title: A Multi-center,Randomized,Double-blind,Placebo,Parallel-controlled Phase II Clinical Study of Jaktinib Hydrochloride Tablets in the Treatment of Moderate and Severe Atopic Dermatitis Patients
Brief Title: Clinical Study of Jaktinib in the Treatment of Patients With Moderate and Severe Atopic Dermatitis
Acronym: AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK011
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Jaktinib 50mg Bid (Experimental): Jaktinib 50mg Bid+ Placebo 50mg Bid+Placebo 75mg Bid
  Interventions: Drug: Jaktinib
- Jaktinib 75mg Bid (Experimental): Jaktinib 75mg Bid+ Placebo 100mg Bid
  Interventions: Drug: Jaktinib
- Jaktinib 100mg Bid (Experimental): Jaktinib 100mg Bid+ Placebo 75mg Bid
  Interventions: Drug: Jaktinib
- placebo (Placebo Comparator): Placebo 100mg Bid+ Placebo 75mg Bid
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Jaktinib — In the morning: 1 tablet of 50mg and 75mg placebo, 1 tablet of 50mg Jaktinib; In the evening: 1 tablet of 50mg and 75mg placebo, 1 tablet of 50mg Jaktinib.
  Arms: Jaktinib 50mg Bid
Drug: Jaktinib — In the morning: 2 tablet of 50mg placebo, 1 tablet of 75mg Jaktinib; In the evening: 2 tablet of 50mg placebo, 1 tablet of 75mg Jaktinib.
  Arms: Jaktinib 75mg Bid
Drug: Jaktinib — In the morning: 1 tablet of 75mg placebo, 2 tablet of 50mg Jaktinib; In the evening: 1 tablet of 75mg placebo, 2 tablet of 50mg Jaktinib.
  Arms: Jaktinib 100mg Bid
Drug: placebo — In the morning: 2 tablet of 50mg placebo, 1 tablet of 75mg placebo;In the evening: 2 tablet of 50mg placebo, 1 tablet of 75mg placebo.
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Jaktinib in participants with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
The study is divided into two stages, the first stage test (1-12 weeks): the main test; the second stage test (13-24 weeks): the extended test.

The main test：The trial set up 4 treatment groups, including 3 dose exploration groups, Jaktinib 50mg Bid, 75mg Bid, 100mg Bid group and 1 placebo control group.

The extended test：Subjects in the placebo group were randomly assigned to receive Jaktinib 50mg Bid, 75mg Bid, and 100mg Bid treatments at a ratio of 1:1:1 (randomized in a blinded state and completed by IWRS in the background), the main test group (50mg Bid, 75mg Bid, 100mg Bid group) subjects still maintain the original dose after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Chinese diagnostic criteria for atopic dermatitis (Zhang's criteria) and be diagnosed as atopic dermatitis.
* Participants must have moderate to severe AD at screening and randomization.
* Participants must have inadequate response to topical medications within 6 months of screening.
* Agree to use emollients daily

Exclusion Criteria:

* Received prior treatment with any oral Janus kinase (JAK) inhibitor less than 4 weeks prior to randomization.
* Have received certain types of vaccinations.
* Participants who do not agree to use adequate contraception during the trial and within 4 weeks after the last dose.
* Any Participants whom the investigator deems inappropriate for participation in this clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving at least a 50% Reduction in Eczema Area and Severity Index (EASI 50) from Baseline | At Week 12
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of atopic dermatitis (AD)

SECONDARY OUTCOMES:
Percentage of Participants Achieving IGA of 0 or 1. | Treatment at 2,4,8,12,16,20,24 weeks
  The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1 with a ≥2 Point Improvement | Treatment at 2,4,8,12,16,20,24 weeks
  The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, Principal Investigator — Central South University
Locations (1):
- The second xiangya hospital of central south university, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No